CLINICAL TRIAL: NCT02469311
Title: Prospective, Randomized Study Evaluating The Efficacy of Chlorhexidine Gluconate Impregnated No-Rinse Cloths in Reducing Surgical Site Infections for Total Hip and Knee Arthroplasty.
Brief Title: Prospective, Randomized Study Evaluating The Efficacy of Chlorhexidine Gluconate Impregnated No-Rinse Cloths.
Acronym: SAGE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary results showed that the use of the cloths helped prevent infections.
Sponsor: LifeBridge Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LifeBridgeH
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis; Infection
Keywords: infection; arthroplasty; chlorhexidine; hip; knee
MeSH Terms: conditions — Osteoarthritis; Infections | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Primary Control TKA (Sham Comparator): Patients undergoing a first or primary total knee arthroplasty will be randomized to the intervention of Standard of care bathing with antibacterial soap and water.
  Interventions: Other: Standard of care bathing with antibacterial soap and water
- Primary Treatment TKA (Active Comparator): Patients undergoing a first or primary total knee arthroplasty will be randomized to the intervention of chlorhexidine impregnated cloths.
  Interventions: Other: chlorhexidine impregnated cloths
- Revision Treatment TKA (Active Comparator): Patients undergoing a second or subsequent or a revision total knee arthroplasty will be randomized to the intervention of a chlorhexidine impregnated cloths.
  Interventions: Other: chlorhexidine impregnated cloths
- Revision Control TKA (Sham Comparator): Patients undergoing a second or revision total knee arthroplasty will be randomized to the intervention of Standard of care bathing with antibacterial soap and water.
  Interventions: Other: Standard of care bathing with antibacterial soap and water
- Primary Control THA (Sham Comparator): Patients undergoing a first or primary total hip arthroplasty will be randomized to the intervention of Standard of care bathing with antibacterial soap and water.
  Interventions: Other: Standard of care bathing with antibacterial soap and water
- Primary Treatment THA (Active Comparator): Patients undergoing a first or primary total hip arthroplasty will be randomized to the intervention of chlorhexidine impregnated cloths.
  Interventions: Other: chlorhexidine impregnated cloths
- Revision Control THA (Sham Comparator): Patients undergoing a second or revision total hip arthroplasty will be randomized to the intervention of Standard of care bathing with antibacterial soap and water.
  Interventions: Other: Standard of care bathing with antibacterial soap and water
- Revision Treatment THA (Active Comparator): Patients undergoing a second or subsequent or a revision total knee arthroplasty will be randomized to the intervention of chlorhexidine impregnated cloths.
  Interventions: Other: chlorhexidine impregnated cloths

INTERVENTIONS:
Other: chlorhexidine impregnated cloths — Pre-operative use of Chlorhexidine cloths night before and morning of surgery
  Arms: Primary Treatment THA; Primary Treatment TKA; Revision Treatment THA; Revision Treatment TKA
Other: Standard of care bathing with antibacterial soap and water — Patients had standard pre-operative bathing with antibacterial soap and water the night before surgery.
  Arms: Primary Control THA; Primary Control TKA; Revision Control THA; Revision Control TKA

SUMMARY:
Subjects in the study were randomized to a treatment group using Chlorhexidine cloths or a standard-of-care group who only had a bath with antibacterial soap and water. Both groups received standard infection control practices during admission.

DETAILED DESCRIPTION:
Between March 2012 and November 2012, patients scheduled for total hip arthroplasty (THA) or total knee arthroplasty (TKA) were randomized (539 patients; 554 arthroplasties) at the time of their preoperative clinic visit. Patients in the chlorhexidine protocol group (275 arthroplasties) applied 2% chlorhexidine gluconate-impregnated cloths to their skin the night before and the morning of surgical admission. Patients in the standard of care group (279 arthroplasties) took a bath with soap and water the night before surgical admission. Both groups were subject to standard infection control practices during admission. The primary outcome was periprosthetic infection incidence within one year of surgery, and secondary outcomes included the potential influence of risk factors for periprosthetic infection and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Joint replacement surgery for any reason
* 18 years or older

Exclusion Criteria:

* unable to comply with study requirements
* were pregnant
* were under the age of 18 years
* medical history of immunosuppression or systemic disease e.g. human immunodeficiency virus, status-post organ transplantation
* received greater than 10 milligrams of prednisone equivalent for more than 10 days within 90 days prior to enrollment;
* chronic hepatitis B or C infection
* had an infection in or around the joint requiring surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The incidence of periprosthetic infection. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mont, MD, Principal Investigator — Director, Rubin Instituted for Advanced Orthopedics and Joint Preservation and Replacement